CLINICAL TRIAL: NCT04929015
Title: Peritoneal Carcinomatosis Leveraging ctDNA Guided Treatment in GI Cancer Study (PERICLES Study)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Henry Richard Alexander, MD, Chief Surgical Officer, Rutgers Cancer Institute of New Jersey, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro2021000017; 072013 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH); NCI-2021-02123 (Registry Identifier: NCI CTRP registry)
Record Dates: First submitted 2021-05-31; First posted 2021-06-18 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Appendix Carcinoma by AJCC V8 Stage; Colorectal Carcinoma by AJCC V8 Stage; Digestive System Neoplasm; Esophageal Carcinoma by AJCC V8 Stage; Gastric Carcinoma by AJCC V8 Stage; Liver and Intrahepatic Bile Duct Carcinoma; Peritoneal Carcinomatosis
MeSH Terms: conditions — Digestive System Neoplasms; Carcinoma, Hepatocellular; Peritoneal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic (biospecimen collection) (Experimental): Patients will receive standard treatment with surgery, HIPEC, and chemotherapy as appropriate to the patient situation, extent of disease and multi-disciplinary evaluation.
  Patients undergo blood sample collection for ctDNA analysis at baseline, pre-surgery, post-surgery and every 3 months up to 2 years.
  Patients undergo tissue collection before or during surgery and their medical records are reviewed.
  Interventions: Procedure: Biospecimen Collection - blood and tissue sample collection; Other: Electronic Health Record Review

INTERVENTIONS:
Procedure: Biospecimen Collection - blood and tissue sample collection — The original tissue sample from each patient will be obtained at time of surgery or prior to surgery. Plasma for ctDNA will be obtained at baseline, pre-surgery, post-surgery and every 3 months up 2 years
Other: Electronic Health Record Review — Medical record reviewed

SUMMARY:
This clinical trial collects biospecimen samples to create a personalized ctDNA test to guide treatment for patients with gastrointestinal cancer with peritoneal carcinomatosis. Deoxyribonucleic acid, or DNA, is the material that carries all the information about how a living thing will work and function. Everyone is born with the same DNA in all our cells throughout our body. Sometimes, some of the cells in the body develop abnormalities in the DNA that cause those cells to grow abnormally and uncontrollably. Cancer occurs when there is abnormal and uncontrolled growth of cells. The DNA in cancer cells is therefore different from the DNA someone is born with. The Signatera ctDNA assay is a laboratory test that takes tumor (cancer) tissue and evaluates it for unique tumor DNA. This evaluation is used to create a report (otherwise known as an assay) personalized to each person's cancer. The personalized assay creates a personalized blood test to detect the level of abnormal DNA from the cancer that may be circulating in the body. Once this personalized blood assay is designed, it may be used to monitor a person's blood for the presence of ctDNA, which will indicate the presence or absence of cancer over time, even after treatment.

DETAILED DESCRIPTION:
This study is an exploratory analysis of the utility of ctDNA as a sensitive biomarker in patients with Peritoneal Carcinomatosis treated with chemotherapy, CRS and/or hyperthermic intraperitoneal chemotherapy (HIPEC).

OBJECTIVES:

I. To measure changes in circulating tumor deoxyribonucleic acid (ctDNA) in patients with peritoneal carcinomatosis (PC) from gastrointestinal (GI) cancers who are candidates for cytoreductive surgery (CRS) with or without hyperthermic intraperitoneal chemotherapy (HIPEC).

II. To determine the percentage of patients on protocol with undetectable ctDNA (clearance rate) after complete CRS.

III. To identify any associations between clinical staging of CRS and measurable ctDNA.

IV. To assess changes in ctDNA levels in response to chemotherapy in patients with PC.

V. To guide treatment based on ctDNA response.

OUTLINE:

Patients may receive induction chemotherapy at the discretion of the treating physician for up to 6 months. Patients undergo blood sample collection for ctDNA analysis at baseline, post chemotherapy/pre-surgery, 3-4 weeks post CRS/HIPEC, then every 3 months over 2 years. Patients also undergo tissue collection before or during surgery and their medical records are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed carcinoma of presumed gastrointestinal origin (gastric, esophageal, colorectal, appendiceal, hepatobiliary or peritoneal carcinomatosis of apparent GI primary) with documented diffuse peritoneal carcinomatosis, either by conventional imaging studies, positive ascitic fluid analysis, or surgical staging
* Measurable or evaluable disease by cross-sectional imaging studies
* Patients must be candidates for possible surgical cytoreduction (with or without HIPEC) as determined by a study surgical oncologist
* Age >= 18 years
* Estimated life expectancy of at least 12 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Patients must sign informed consent
* Be willing to present for medical exams, blood draws and imaging as scheduled in protocol
* Be able to donate two 10 mL tubes of blood every 3 months
* Women of childbearing potential will undergo routine screening evaluation for pregnancy prior to enrollment and be managed per standard of care

Exclusion Criteria:

* Patients without a confirmed pathologic diagnosis of carcinoma
* Second uncontrolled primary malignancy
* Patients who are pregnant
* Patients who cannot undergo a therapeutic surgical cytoreduction
* Bone marrow transplant or other organ transplant recipient
* Any unstable, serious co-existing medical conditions including but not limited to myocardial infarction, coronary bypass surgery, unstable angina, cardiac arrhythmias, clinically evident congestive heart failure, or cerebrovascular accident within 6 months prior to screening
* Patients with cardiovascular or pulmonary risk factors contributing to high risk for surgical complications, at the discretion of the surgeon
* Serious concomitant systemic disorder that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-04-29 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Clearance rate of circulating tumor deoxyribonucleic acid (ctDNA) with cytoreductive surgery (CRS) | Baseline, pre-surgery, 3- 4 weeks post-surgery and then every 3 months up to 2 years after cytoreductive surgery (CRS)
  Will compare results with clinical staging of CRS (surgical staging, surgical outcomes, Peritoneal Carcinoma Index [PCI] and cytoreduction [CC] score). ctDNA clearance rate defined as the % of patients on our protocol with undetectable ctDNA. Will associate ctDNA changes with clinical response by Response Evaluation Criteria in Solid Tumors and surgical staging, surgical outcomes, PCI and CC score using standard T-testing, log-rank analysis or similar non-parametric testing.
Correlation of ctDNA clearance with activity of chemotherapy | Baseline, pre-surgery, 3-4 weekd post-surgery and then every 3 months up to 2 years after cytoreductive surgery (CRS)
  Will correlate ctDNA clearance with activity of chemotherapy in this disease pre-op and post-op

SECONDARY OUTCOMES:
Positivity rate of ctDNA in patients with peritoneal carcinomatosis | Baseline, pre-surgery, 3-4 weeks post-surgery and then every 3 months up to 2 years after cytoreductive surgery (CRS)
  ctDNA will be obtained at baseline, pre-surgery, post-surgery and every 3 months up to 2 years
ctDNA and its association with results of next generation sequence (NSG) analysis from original tumor tissue. | Baseline, pre-surgery, 3-4 weeks post-surgery and then every 3 months up to 2 years after cytoreductive surgery (CRS)
  ctDNA will be obtained at baseline, pre-surgery, 3-4 weeks post-surgery and then every 3 months up to 2 years. ctDNA from blood samples will be compared with the results of NSG analysis from original tumor tissue
Associations between CEA levels and ctDNA levels | Baseline, pre-surgery, 3-4 weeks post-surgery and every 3 months up to 2 years after cytoreductive surgery (CRS)
  ctDNA will be obtained at baseline, pre-surgery, post-surgery and every 3 months up to 2 years
Associations between CA19.9 levels and ctDNA levels | Baseline, pre-surgery, 3-4 weeks post-surgery and every 3 months up to 2 years after cytoreductive surgery (CRS)
  ctDNA will be obtained at baseline, pre-surgery, post-surgery and every 3 months up to 2 years
Associations between CA125 levels and ctDNA levels | Baseline, pre-surgery, 3-4 weeks post-surgery and every 3 months up to 2 years after cytoreductive surgery (CRS)
  ctDNA will be obtained at baseline, pre-surgery, post-surgery and every 3 months up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry R Alexander, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (2):
- United States (2):
  - RWJBarnabas Health - Cooperman Barnabas, Livingston, Livingston, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey

IPD SHARING:
Plan to Share IPD: No